CLINICAL TRIAL: NCT01000311
Title: A Phase 3, Randomized, Open Label, Controlled Multicenter Study to Evaluate the Safety and Immunogenicity of 4 Doses of MenACWY Conjugate Vaccine, Administered Concomitantly With Routine Vaccines, Among Infants Aged 2 Months
Brief Title: A Study to Evaluate the Safety and Immunogenicity of 4 Doses of MenACWY Conjugate Vaccine, Administered Concomitantly With Routine Vaccines, Among Infants Aged 2 Months
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Vaccines (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: V59_33
Record Dates: First submitted 2009-10-22; First posted 2009-10-23 (Estimated); Results first posted 2014-03-26 (Estimated); Last update posted 2014-04-21 (Estimated); Status verified 2014-04

CONDITIONS: Meningococcal Disease
Keywords: MenACWY conjugate vaccine in infants; Meningococcal vaccine in infants; MenACWY
MeSH Terms: conditions — Meningococcal Infections | interventions — MenACWY-CRM vaccine; diphtheria-tetanus-five component acellular pertussis-inactivated poliomyelitis -Haemophilus influenzae type b conjugate vaccine; Tetanus Toxoid; pentacel; Hepatitis B Vaccines; Engerix-B; Heptavalent Pneumococcal Conjugate Vaccine; 13-valent pneumococcal vaccine; Rubella Vaccine; Measles-Mumps-Rubella Vaccine

ARMS (2):
- MenACWY-CRM + Routine Vaccines (Experimental): Infants received 3 doses of MenACWY-CRM at 2, 4 and 6 months as a infant series vaccination and a toddler dose at 12 months of age.
  Infants also received routine vaccines - 3 doses each of DTaP-IPV/Hib, HBV and PCV at 2, 4 and 6 months; and 1 dose each of PCV and MMR at 12 months.
  Interventions: Biological: MenACWY-CRM; Biological: DTaP-IPV/Hib; Biological: HBV; Biological: PCV; Biological: MMR
- Routine Vaccines (Experimental): Infants received routine vaccines - 3 doses each of DTaP-IPV/Hib, HBV and PCV at 2, 4 and 6 months; and 1 dose each of PCV and MMR at 12 months.
  In addition subjects were offered a dose of MenACWY-CRM at 18 months as a benefit of participating in this study. However, blood was not drawn for immunogenicity analysis after this dose.
  Interventions: Biological: DTaP-IPV/Hib; Biological: HBV; Biological: PCV; Biological: MMR

INTERVENTIONS:
Biological: MenACWY-CRM — One dose (0.5 mL) of MenACWY conjugate vaccine supplied as an extemporaneous mixing just before injection of the lyophilized component (MenA) reconstituted with the liquid component (MenCWY) was administered at 2, 4, 6 and 12 months of age as IM injections in the anterolateral area of the thigh.
  Arms: MenACWY-CRM + Routine Vaccines
Biological: DTaP-IPV/Hib — IM injections of 3 doses of 0.5 mL each of DTaP-IPV/Hib supplied in prefilled vial were administered at 2, 4 and 6 months of age in the anterolateral area of the thigh.
  Other Names: Combined diphtheria, tetanus toxoid, acellular pertussis and inactivated polio vaccine containing Haemophilus influenzae type B vaccine; Pentacel
Biological: HBV — IM injections of 3 doses of 0.5 mL each of HBV supplied in prefilled vial were administered at 2, 4 and 6 months of age in the anterolateral area of the thigh.
  Other Names: Hepatitis B virus vaccine; Engerix-B
Biological: PCV — IM injections of 4 doses of 0.5 mL each of PCV supplied in prefilled vial were administered at 2, 4, 6 and 12 months of age in the anterolateral area of the thigh.
  Other Names: Heptavalent Streptococcus pneumonia vaccine; Prevnar (PCV-7); Prevnar 13 (PCV-13)
Biological: MMR — Subcutaneous (SC) injection of 1 dose of 0.5 mL of MMR obtained by extemporaneous mixing just before injection of powder and the solvent for solution was administered at 12 months of age in the anterolateral area of the thigh.
  Other Names: Measles, mumps, and rubella vaccine; M-M-R II

SUMMARY:
This Phase 3 study is designed to demonstrate the safety and immunogenicity of MenACWY and non-interference of concomitant routine vaccines by MenACWY in an infant age group.

ELIGIBILITY:
Inclusion Criteria:

1. Two month-old infants, born after a full-term pregnancy with an estimated gestational age ≥37 weeks and a birth weight ≥2.5 kg.
2. Documented written informed consent provided by the parent/legal representative after the nature of the study had been explained.
3. Parent/legal representative was available for all visits scheduled in the study.
4. Subjects were in good health as determined by:

   1. medical history
   2. physical assessment
   3. clinical judgment of the investigator

Exclusion Criteria:

1. Subjects who previously received any meningococcal vaccines or vaccines against diphtheria, tetanus, pertussis, polio (IPV or OPV), H. influenzae type b (Hib) or pneumococcus. Exceptions: prior doses HBV vaccination (one or two doses) are permitted.
2. Subjects who had a previous confirmed or suspected disease caused by N. meningitidis, C. diphtheriae, C. tetani, poliovirus, Hepatitis B, Hib, pneumococcus or B. pertussis (history of laboratory confirmed, or clinical condition of paroxysmal cough for a period of longer than or equal to 2 weeks associated with apnea or whooping).
3. Subjects who had household contact with and/or intimate exposure to an individual with laboratory confirmed N. meningitidis, B. pertussis, Hib, C. diphtheriae, polio, or pneumococcal infection at any time since birth.
4. Subjects who had a history of anaphylactic shock, asthma, urticaria or other allergic reaction after previous vaccinations or known hypersensitivity to any vaccine component.
5. Subjects who had experienced significant acute or chronic infection within the previous 7 days or have experienced fever (temperature ≥ 38.0°C [100.4°F]) within the previous 3 days.
6. Subjects who had any serious acute or chronic disease, neurological disease including seizures, congenital defects, or cytogenic disorders (e.g., Down syndrome).
7. Subjects who had a known or suspected autoimmune disease or persistent impairment/alteration of immune function.
8. Subjects who had a suspected or known HIV infection or were born to a mother known to be HIV positive.
9. Subjects who had ever received blood, blood products and/or plasma derivatives or any parenteral immunoglobulin preparation (including Hepatitis B immune globulin).
10. Subjects who had a known bleeding diathesis, or any condition that may be associated with a prolonged bleeding time.
11. Subjects who with their parents/legal representatives were planning to leave the area of the study site before the end of the study period.
12. Subjects who had any condition which, in the opinion of the investigator, might interfere with the evaluation of the study objectives.
13. Subjects who received any investigational agents or vaccines since birth or who expect to receive an investigational agent or vaccine prior to the completion of the study.
14. Subjects who were relatives of site research staff working on this study.

Ages: 55 Days to 89 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 529 (Actual)
Dates: Start 2009-11; Primary Completion 2011-11 (Actual); Study Completion 2011-11 (Actual)

CONTACTS AND LOCATIONS:
Locations (46):
- United States (42):
  - 37 Alabama Clinical Therapeutics LLC 52 Medical Park East Drive Suite 203, Birmingham, Alabama
  - 15 Northwest Arkansas Pediatric Clinic 3383 N. Mana Court Suite 101, Fayetteville, Arkansas
  - 6 Children's Clinic of Jonesboro AR 800 South Church Street Suite 400 and 204, Jonesboro, Arkansas
  - 9 San Fernando Valley Research Associates 7111 Winnetka Avenue Suite 14, Canoga Park, California
  - 17 Edinger Medical Group Research Center 9900 Talbert Avenue Suite 204, Fountain Valley, California
  - 28 Madera Family Medical Group 1111 West 4th Street, Madera, California
  - 38 Center for Clinical Trials LLC 16660 Paramount Blvd Suite 301, Paramount, California
  - 8 Pharmax Research Clinic 7200 NW 7th Street Suite 350, Miami, Florida
  - 48 Cotton O'Neil Clinical Research Center 4100 SW 15th Street, Topeka, Kansas
  - 47 Cotton O'Neil Clinical Research Center 6725 SW 29th Street, Topeka, Kansas
  - 29 Kentucky Pediatric/Adult Research 201 South 5th Street, Bardstown, Kentucky
  - 4 Nassim McMonigle Mescia and Associates 5512 Bardstown Road Suite 2, Louisville, Kentucky
  - 40 Brownsboro Park Pediatrics 5512 Bardstown Road Suite 2, Louisville, Kentucky
  - 24 University Of Louisville 555 South Floyd Street, Louisville, Kentucky
  - 26 University Of Louisville 230 East Broadway, Louisville, Kentucky
  - 30 Kentucky Pediatric/Adult Research 102 West Depot Street, Springfield, Kentucky
  - 27 Ark-La-Tex Children's Clinic 1025 Highway 80 E, Haughton, Louisiana
  - 13 Willis Knighton Physician Network- Portico Pediatrics 7847 Youree Drive, Shreveport, Louisiana
  - 35 Southwestern Medical Clinic P.C. 2002 S 11th Street, Niles, Michigan
  - 25 Center for Pharmaceutical Research 1010 Carondelet Drive Suite 426, Kansas City, Missouri
  - 31 Senders Pediatrics 2054 South Green Road, Cleveland, Ohio
  - 5 Dayton Clinical Research 1100 Salem Ave., Dayton, Ohio
  - 14 Ohio Pediatrics Research Association 7371 Brandt Pike Suite C, Huber Heights, Ohio
  - 22 Ohio Pediatrics Research Association 1775 Delco Park Drive, Kettering, Ohio
  - 45 Oklahoma State University Physicians 635 W 11th St, Tulsa, Oklahoma
  - 33 Primary Physicians Research Inc. 1580 McLaughlin Run Road, Pittsburgh, Pennsylvania
  - 34 Primary Physicians Research Inc. 1580 McLaughlin Run Road, Pittsburgh, Pennsylvania
  - 10 Holston Medical Group 105 W. Stone Drive Suite 3B, Kingsport, Tennessee
  - 23 Focus Research Group 201 Signature Place, Lebanon, Tennessee
  - 7 Amarillo Children's Clinical Research #17 Care Circle, Amarillo, Texas
  - 46 Pediatric Healthcare of Northwest Houston P.A. 12015 Louetta Road Suite 100, Houston, Texas
  - 12 Pediatric Healthcare of Northwest Houston P.A. 13406 Medical Complex Drive Suite 200, Tomball, Texas
  - 16 Westside Medical 1477 North 2000 West, Clinton, Utah
  - 42 Wee Care Pediatrics 934 S. Main Street Suite 8, Layton, Utah
  - 43 Wee Care Pediatrics 1580 W. Antelope Drive Suite 100, Layton, Utah
  - 19 Pediatric Care 1675 North Freedom Blvd Building 3, Provo, Utah
  - 44 Wee Care Pediatrics 5991 S. 3500 W Suite 100 Rock Run Plaza, Roy, Utah
  - 18 Copperview Medical Center 3556 West 9800 South, South Jordan, Utah
  - 39 Dixie Pediatrics 1240 E 100 S Suite 14, St. George, Utah
  - 41 Wee Care Pediatrics 1792 W. 1700 S. Suite 102, Syracuse, Utah
  - 36 Dominion Medical Associates 304 East Leigh Street, Richmond, Virginia
  - 21 CAMC Health Education and Research Institute 3100 McCorkle Ave. S.E. Suite 806, Charleston, West Virginia
- Australia (3):
  - 3 Sydney Children's Hospital Strasser Lab. Level 3 High Street, Randwick, New South Wales
  - 2 Royal Children's Hospital Herston Road, Herston, Queensland
  - 1 Murdoch Childrens Research Institute C/- School of Population Health The University of Melbourne, Carlton, Victoria
- 20 Medicor Research Inc 359 Riverside Suite 200, Greater Sudbury, Ontario, Canada

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were enrolled at 42 study sites in the United States, 3 sites in Australia and 1 site in Canada.
Pre-assignment Details: All enrolled subjects were included in the study.
Groups:
- MenACWY-CRM + Routine Vaccines: Infants received 3 doses of MenACWY-CRM at 2, 4 and 6 months as a infant series vaccination and a toddler dose at 12 months.
  Infants also received routine vaccines - 3 doses each of DTaP-IPV/Hib, HBV and PCV at 2, 4 and 6 months; and 1 dose each of PCV and MMR at 12 months.
- Routine Vaccines: Infants received routine vaccines - 3 doses each of DTaP-IPV/Hib, HBV and PCV at 2, 4 and 6 months; and 1 dose each of PCV and MMR at 12 months.
Period: Overall Study
Arm/Group | MenACWY-CRM + Routine Vaccines | Routine Vaccines
Started | 258 | 271
Completed | 213 | 201
Not Completed | 45 | 70
Not completed — Adverse Event | 2 | 5
Not completed — Withdrawal by Subject | 16 | 24
Not completed — Lost to Follow-up | 15 | 24
Not completed — Protocol Violation | 1 | 2
Not completed — Inappropriate enrollment | 2 | 0
Not completed — Administrative reason | 9 | 15

BASELINE CHARACTERISTICS:
Population: Analysis was performed on all enrolled subjects.
Groups:
- Total: Total of all reporting groups
Arm/Group | MenACWY-CRM + Routine Vaccines | Routine Vaccines | Total
Number analyzed (Participants) | 258 | 271 | 529
Age, Continuous [Mean (Standard Deviation); unit: Days] | 64.7 (6.5) | 65.4 (7.4) | 65.1 (7.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 125 | 130 | 255
  Male | 133 | 141 | 274

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Subjects With hSBA Titer ≥1:8 Against Serogroup A, C, W and Y One Month After Toddler Vaccination of MenACWY-CRM
Description: Immunogenicity was measured as the percentage of subjects who achieved hSBA titer ≥1:8 against meningococcal serogroup A, C, W and Y, evaluated by serum bactericidal assay using human complement (hSBA), at baseline and one month after toddler dose of MenACWY-CRM administered at 12 months of age.
  The immune response was considered sufficient if the lower limit of the two-sided 95% confidence intervals (CIs) for the percentage of subjects with hSBA titer ≥1:8, at one month after toddler vaccination, was greater than 85% for the serogroup C, W, or Y and greater than 80% for the serogroup A.
Time Frame: Baseline and one month after fourth-dose of MenACWY-CRM
Population: Analysis was done on the per-protocol (PP) toddler dataset for MenACWY-CRM, i.e. the subjects who received all the relevant doses of vaccine correctly; provided evaluable serum samples at the relevant time points; and had no major protocol violation as defined prior to database lock.
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | MenACWY-CRM + Routine Vaccines | Routine Vaccines
Number analyzed (Participants) | 170 | 178
Percentage of subjects
  Serogroup A - Baseline (N=170,178) | 2 [0 to 5] | 1 [0.014 to 3]
  Serogroup A - Post-4th dose (N=168,175) | 89 [83 to 93] | 2 [0 to 5]
  Serogroup C - Baseline (N=166,174) | 7 [3 to 12] | 7 [4 to 12]
  Serogroup C - Post-4th dose (N=156,171) | 95 [90 to 98] | 2 [1 to 6]
  Serogroup W - Baseline (N=152,164) | 13 [8 to 20] | 15 [10 to 21]
  Serogroup W - Post-4th dose (N=153,165) | 97 [93 to 99] | 7 [3 to 12]
  Serogroup Y - Baseline (N=144,150) | 8 [4 to 13] | 4 [1 to 9]
  Serogroup Y - Post-4th dose (N=153,159) | 96 [92 to 99] | 1 [0 to 4]
Statistical Analysis 1: Comparison: MenACWY-CRM + Routine Vaccines; The null hypothesis associated with the primary objective was that the immune response was considered sufficient if the lower limit of the two-sided 95% confidence intervals (CIs) for the percentage of subjects with hSBA titer ≥1:8, at one month after 4th dose was greater than 80% for the serogroup A; Test type: Superiority or Other; Lower limit of 95% confidence interval = 83, 95% CI 2-sided [83 to 93]
Statistical Analysis 2: Comparison: MenACWY-CRM + Routine Vaccines; The null hypothesis associated with the primary objective was that the immune response was considered sufficient if the lower limit of the two-sided 95% CI for the percentage of subjects with hSBA titer ≥1:8, at one month after 4th dose was greater than 85% for the serogroup C; Test type: Superiority or Other; Lower limit of 95% confidence interval = 90, 95% CI 2-sided [90 to 98]
Statistical Analysis 3: Comparison: MenACWY-CRM + Routine Vaccines; The null hypothesis associated with the primary objective was that the immune response was considered sufficient if the lower limit of the two-sided 95% CI for the percentage of subjects with hSBA titer ≥1:8, at one month after 4th dose was greater than 85% for the serogroup W; Test type: Superiority or Other; Lower limit of 95% confidence interval = 93, 95% CI 2-sided [93 to 99]
Statistical Analysis 4: Comparison: MenACWY-CRM + Routine Vaccines; The null hypothesis associated with the primary objective was that the immune response was considered sufficient if the lower limit of the two-sided 95% CI for the percentage of subjects with hSBA titer ≥1:8, at one month after 4th dose was greater than 85% for the serogroup Y; Test type: Superiority or Other; Lowe limit of 95% confidence interval = 92, 95% CI 2-sided [92 to 99]

2. Secondary Outcome: hSBA Geometric Mean Titers Against Serogroup A, C, W and Y One Month After Toddler Vaccination of MenACWY-CRM
Description: Immunogenicity was measured as the hSBA geometric mean titers (GMTs) directed against meningococcal serogroup A, C, W and Y, at baseline and one month after toddler dose of MenACWY-CRM administered at 12 months of age.
Time Frame: Baseline and one month after fourth-dose of MenACWY-CRM
Population: Analysis was performed on the PP toddler dataset for MenACWY-CRM vaccination.
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | MenACWY-CRM + Routine Vaccines | Routine Vaccines
Number analyzed (Participants) | 168 | 175
Titers
  Serogroup A - Baseline (N=139,145) | 2.07 [1.98 to 2.16] | 2.01 [1.99 to 2.03]
  Serogroup A - Post-4th dose (N=168,175) | 54 [44 to 67] | 1.87 [1.55 to 2.27]
  Serogroup C - Baseline (N=126,136) | 2.49 [2.2 to 2.83] | 2.44 [2.2 to 2.7]
  Serogroup C - Post-4th dose (N=156,171) | 135 [107 to 171] | 1.94 [1.56 to 2.4]
  Serogroup W - Baseline (N=113,126) | 2.99 [2.49 to 3.6] | 2.97 [2.52 to 3.51]
  Serogroup W - Post-4th dose (N=153,165) | 215 [167 to 277] | 2.15 [1.77 to 2.6]
  Serogroup Y - Baseline (N=108,113) | 2.43 [2.19 to 2.71] | 2.32 [2.13 to 2.52]
  Serogroup Y - Post-4th dose (N=153,159) | 185 [148 to 233] | 1.89 [1.56 to 2.29]

3. Secondary Outcome: Percentage of Subjects With hSBA Titers ≥1:8, and Four-Fold Increase in hSBA Titers Against Serogroup A, C, W and Y One Month After Three Dose Infant Series Vaccination of MenACWY-CRM
Description: Immunogenicity was measured as the percentage of subjects with hSBA titers ≥1:8 against meningococcal serogroup A, C, W and Y, before (baseline) and one month after 3 infant doses of MenACWY-CRM administered at 2, 4 and 6 months of age.
  Percentage of subjects who achieved at least four-fold rise in hSBA titers against serogroup A, C, W and Y was measured one month after 3 infant doses of MenACWY-CRM.
Time Frame: Baseline and one month after third infant dose of MenACWY-CRM
Population: Analysis was performed on the PP dataset of MenACWY-CRM infant vaccination series.
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | MenACWY-CRM + Routine Vaccines | Routine Vaccines
Number analyzed (Participants) | 202 | 208
Percentage of subjects
  Serogroup A - hSBA ≥1:8-Baseline (N=170,178) | 2 [0 to 5] | 1 [0.014 to 3]
  Serogroup A - hSBA ≥1:8 -Post-3rd dose(N=202,208) | 76 [69 to 81] | 1 [0 to 4]
  Serogroup C - hSBA ≥1:8 -Baseline(N=166,174) | 7 [3 to 12] | 7 [4 to 12]
  Serogroup C - hSBA ≥1:8 -Post-3rd dose(N=199,206) | 94 [90 to 97] | 1 [0 to 4]
  Serogroup W - hSBA ≥1:8 -Baseline(N=152,164) | 13 [8 to 20] | 15 [10 to 21]
  Serogroup W - hSBA ≥1:8 -Post-3rd dose(N=194,202) | 98 [95 to 99] | 3 [1 to 7]
  Serogroup Y - hSBA ≥1:8 -Baseline(N=144,150) | 8 [4 to 13] | 4 [1 to 9]
  Serogroup Y - hSBA ≥1:8 -Post-3rd dose(N=188,196) | 94 [89 to 97] | 3 [1 to 6]
  Serogroup A - 4-fold rise-Post-3rd dose(N=170,177) | 78 [71 to 84] | 2 [0 to 5]
  Serogroup C - 4-fold rise-Post-3rd dose(N=164,171) | 94 [89 to 97] | 1 [0 to 4]
  Serogroup W - 4-fold rise-Post-3rd dose(N=147,158) | 93 [87 to 96] | 2 [0 to 5]
  Serogroup Y -4-fold rise-Post-3rd dose(N=135,142) | 93 [87 to 96] | 2 [0 to 6]

4. Secondary Outcome: hSBA Geometric Mean Titers Against Serogroup A, C, W and Y One Month After Three Dose Infant Series Vaccination of MenACWY-CRM
Description: Immunogenicity was measured as the hSBA GMTs directed against meningococcal serogroups A, C, W and Y before (baseline) and one month after 3 infants doses of MenACWY-CRM administered at 2, 4 and 6 months of age.
Time Frame: Baseline and one month after third infant dose of MenACWY-CRM
Population: Analysis was performed on the PP dataset of MenACWY-CRM infant vaccination series.
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | MenACWY-CRM + Routine Vaccines | Routine Vaccines
Number analyzed (Participants) | 202 | 209
Titers
  Serogroup A - Baseline (N=170,178) | 2.09 [2 to 2.18] | 2.05 [1.98 to 2.12]
  Serogroup A - Post-3rd dose (N=202,208) | 21 [17 to 26] | 2.08 [1.99 to 2.17]
  Serogroup C - Baseline (N=166,174) | 2.49 [2.25 to 2.76] | 2.39 [2.18 to 2.61]
  Serogroup C - Post-3rd dose (N=199,206) | 74 [62 to 87] | 1.94 [1.64 to 2.3]
  Serogroup W - Baseline (N=152,164) | 2.94 [2.52 to 3.43] | 2.98 [2.58 to 3.45]
  Serogroup W - Post-3rd dose (N=194,202) | 79 [67 to 92] | 1.94 [1.68 to 2.24]
  Serogroup Y - Baseline (N=144,150) | 2.52 [2.28 to 2.77] | 2.26 [2.12 to 2.41]
  Serogroup Y - Post-3rd dose (N=188,196) | 51 [43 to 61] | 2.13 [2.02 to 2.25]

5. Secondary Outcome: Percentage of Subjects With Seroresponse to Routine Concomitant Vaccinations One Month After Infant Series, When Routine Vaccines Are Administered With MenACWY-CRM Compared With When Routine Vaccines Are Given Alone
Description: The immune seroresponse to routine concomitant vaccination was measured as the percentages of subjects with pre-specified cut-off limit of ≥0.1 IU/mL (Diphtheria and Tetanus); ≥0.15 μg/mL (Hib); ≥0.35 μg/mL (Pneumococcal antigens, PnC); and ≥10 mIU/mL (Hepatitis B), evaluated using enzyme-linked immunosorbent assay (ELISA) at one month after 3 doses of infant series vaccination administered at 2, 4 and 6 months of age.
  The immune response to pertussis antigens (PT, FHA, Pertactin, FIM) was measured as percentage of subjects with seroresponse (in initially seronegative infants, ≥4 times the lower limit of quantification (LLQ); in initially seropositive infants, at least 4 times prevaccination concentration) by ELISA and percentage of subjects with titer ≥1:8 (Polio types 1, 2, and 3) by neutralization test (NT) one month after 3 doses of infant series vaccination administered at 2, 4 and 6 months of age.
Time Frame: One month after third dose of routine infant series vaccination
Population: Analysis was performed on the PP concomitant, pertussis and hepatitis B infant populations.
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | MenACWY-CRM + Routine Vaccines | Routine Vaccines
Number analyzed (Participants) | 207 | 218
Percentage of subjects
  Diphtheria (≥0.1 IU/mL) (N=207,218) | 99 [96 to 100] | 99 [96 to 100]
  Tetanus (≥0.1 IU/mL) (N=207,218) | 97 [94 to 99] | 97 [93 to 99]
  PT (N=185,191) | 77 [71 to 83] | 81 [75 to 86]
  FHA (N=185,191) | 70 [63 to 76] | 65 [58 to 72]
  Pertactin (N=185,191) | 73 [66 to 79] | 73 [66 to 79]
  FIM (N=185,191) | 74 [67 to 80] | 76 [69 to 82]
  Polio Type 1 - ≥1:8 (N=115,113) | 99 [95 to 100] | 98 [94 to 100]
  Polio Type 2 - ≥1:8 (N=185,179) | 100 [98 to 100] | 99 [97 to 100]
  Polio Type 3 - ≥1:8 (N=164,162) | 99 [97 to 100] | 100 [98 to 100]
  Hepatitis B - ≥10 mIU/mL (N=138,148) | 96 [92 to 99] | 97 [92 to 99]
  PRP-Hib - ≥0.15 μg/mL (N=187,194) | 95 [90 to 97] | 89 [84 to 93]
  PnC 4 - ≥0.35 μg/mL (N=183,178) | 99 [96 to 100] | 98 [94 to 99]
  PnC 6B - ≥0.35 μg/mL (N=183,178) | 86 [80 to 91] | 90 [84 to 94]
  PnC 9V - ≥0.35 μg/mL (N=183,178) | 91 [86 to 95] | 94 [90 to 97]
  PnC 14 - ≥0.35 μg/mL (N=183,178) | 99 [96 to 100] | 99 [96 to 100]
  PnC 18C - ≥0.35 μg/mL (N=183,178) | 95 [90 to 97] | 97 [94 to 99]
  PnC 19F - ≥0.35 μg/mL (N=183,178) | 100 [98 to 100] | 97 [93 to 99]
  PnC 23F - ≥0.35 μg/mL (N=183,178) | 89 [83 to 89] | 94 [89 to 97]
Statistical Analysis 1: Comparison: MenACWY-CRM + Routine Vaccines vs Routine Vaccines; To demonstrate the non-inferiority of seroresponse to diphtheria toxin, when DTaP vaccine is given with MenACWY-CRM compared with when DTaP vaccine is given alone; Test type: Non-Inferiority or Equivalence — The immune seroresponse to diphtheria toxin, when DTaP is given concomitantly with MenACWY-CRM, was considered non-inferior to that of DTaP given alone, if the lower limit of the two-sided 95% CI for the difference in the percentage of subjects with antibody response was greater than or equal to -10%; Miettinen and Nurminen; Group difference = 0, 95% CI 2-sided [-2.9 to 2.6]
Statistical Analysis 2: Comparison: MenACWY-CRM + Routine Vaccines vs Routine Vaccines; To demonstrate the non-inferiority of seroresponse to tetanus toxin, when DTaP vaccine is given with MenACWY-CRM compared with when DTaP vaccine is given alone; Test type: Non-Inferiority or Equivalence — The immune seroresponse to tetanus toxin, when DTaP is given concomitantly with MenACWY-CRM, was considered non-inferior to that of DTaP given alone, if the lower limit of the two-sided 95% CI for the difference in the percentage of subjects with antibody response was greater than or equal to -10%; Miettinen and Nurminen; Group difference = 0, 95% CI 2-sided [-3.3 to 3.9]
Statistical Analysis 3: Comparison: MenACWY-CRM + Routine Vaccines vs Routine Vaccines; To demonstrate the non-inferiority of seroresponse to pertussis toxin (PT), when DTaP vaccine is given, compared with MenACWY-CRM compared with when DTaP vaccine is given alone; Test type: Non-Inferiority or Equivalence — The immune seroresponse to pertussis toxin (PT), when DTaP is given concomitantly with MenACWY-CRM, was considered non-inferior to that of DTaP given alone, if the lower limit of the two-sided 95% CI for the difference in the percentage of subjects with antibody response was greater than or equal to -10%; Miettinen and Nurminen; Group difference = -4, 95% CI 2-sided [-12.1 to 4.3]
Statistical Analysis 4: Comparison: MenACWY-CRM + Routine Vaccines vs Routine Vaccines; To demonstrate the non-inferiority of seroresponse to pertussis FHA antigen, when DTaP vaccine is given with MenACWY-CRM compared with when DTaP vaccine is given alone; Test type: Non-Inferiority or Equivalence — The immune seroresponse to pertussis (FHA antigen), when DTaP is given concomitantly with MenACWY-CRM, was considered non-inferior to that of DTaP given alone, if the lower limit of the two-sided 95% CI for the difference in the percentage of subjects with antibody response was greater than or equal to -10%; Miettinen and Nurminen; Group difference = 4, 95% CI 2-sided [-5.1 to 13.6]
Statistical Analysis 5: Comparison: MenACWY-CRM + Routine Vaccines vs Routine Vaccines; To demonstrate the non-inferiority of seroresponse to pertussis pertactin antigen, when DTaP vaccine is given with MenACWY-CRM compared with when DTaP is given alone; Test type: Non-Inferiority or Equivalence — The immune seroresponse to pertussis pertactin antigen, when DTaP vaccine is given concomitantly with MenACWY-CRM, was considered non-inferior to that of DTaP given alone, if the lower limit of the two-sided 95% CI for the difference in the percentage of subjects with antibody response was greater than or equal to -10%; Miettinen and Nurminen; Group difference = 0, 95% CI 2-sided [-8.8 to 9.1]
Statistical Analysis 6: Comparison: MenACWY-CRM + Routine Vaccines vs Routine Vaccines; To demonstrate the non-inferiority of seroresponse to pertussis FIM antigen, when DTaP vaccine is given with MenACWY-CRM compared with when DTaP vaccine is given alone; Test type: Non-Inferiority or Equivalence — The immune seroresponse to pertussis FIM antigen, when DTaP is given concomitantly with MenACWY-CRM, was considered non-inferior to that of DTaP given alone, if the lower limit of the two-sided 95% CI for the difference in the percentage of subjects with antibody response was greater than or equal to -10%; Miettinen and Nurminen; Group difference = -2, 95% CI 2-sided [-10.6 to 6.8]
Statistical Analysis 7: Comparison: MenACWY-CRM + Routine Vaccines vs Routine Vaccines; To demonstrate the non-inferiority of seroresponse to hepatitis B antigen, when hepatitis B vaccine is given with MenACWY-CRM compared with when hepatitis B vaccine is given alone; Test type: Non-Inferiority or Equivalence — The immune seroresponse to hepatitis B, when given concomitantly with MenACWY-CRM, was considered non-inferior to that of hepatitis B vaccine given alone, if the lower limit of the two-sided 95% CI for the difference in the percentage of subjects with antibody response was greater than or equal to -10%; Miettinen and Nurminen; Group difference = 0, 95% CI 2-sided [-5.2 to 4.5]
Statistical Analysis 8: Comparison: MenACWY-CRM + Routine Vaccines vs Routine Vaccines; To demonstrate the non-inferiority of seroresponse to Hib antigen, when Hib vaccine is given with MenACWY-CRM compared with when Hib vaccine is given alone; Test type: Non-Inferiority or Equivalence — The immune seroresponse to Hib vaccine, when given concomitantly with MenACWY-CRM, was considered non-inferior to that of Hib vaccine given alone, if the lower limit of the two-sided 95% CI for the difference in the percentage of subjects with antibody response was greater than or equal to -10%; Miettinen and Nurminen; Group difference = 5, 95% CI 2-sided [0 to 11.2]
Statistical Analysis 9: Comparison: MenACWY-CRM + Routine Vaccines vs Routine Vaccines; To demonstrate the non-inferiority of seroresponse to polio antigen (Type 1), when IPV routine is given with MenACWY-CRM, compared with when IPV is given alone; Test type: Non-Inferiority or Equivalence — The immune seroresponse to polio antigen (Type 1), when IPV is given concomitantly with MenACWY-CRM, was considered non-inferior to that of IPV given alone, if the lower limit of the two-sided 95% CI for the difference in the percentage of subjects with antibody response was greater than or equal to -5%; Miettinen and Nurminen; Group difference = 1, 95% CI 2-sided [-3.1 to 5.4]
Statistical Analysis 10: Comparison: MenACWY-CRM + Routine Vaccines vs Routine Vaccines; To demonstrate the non-inferiority of seroresponse to polio antigen (Type 2), when IPV routine is given with MenACWY-CRM, compared with when IPV is given alone; Test type: Non-Inferiority or Equivalence — The immune seroresponse to polio antigen (Type 2), when IPV is given concomitantly with MenACWY-CRM, was considered non-inferior to that of IPV given alone, if the lower limit of the two-sided 95% CI for the difference in the percentage of subjects with antibody response was greater than or equal to -5%; Miettinen and Nurminen; Group difference = 1, 95% CI 2-sided [-1.4 to 3]
Statistical Analysis 11: Comparison: MenACWY-CRM + Routine Vaccines vs Routine Vaccines; To demonstrate the non-inferiority of seroresponse to polio antigen (Type 3), when IPV routine is given with MenACWY-CRM, compared with when IPV is given alone; Test type: Non-Inferiority or Equivalence — The immune seroresponse to polio antigen (Type 3), when IPV is given concomitantly with MenACWY-CRM, was considered non-inferior to that of IPV given alone, if the lower limit of the two-sided 95% CI for the difference in the percentage of subjects with antibody response was greater than or equal to -5%; Miettinen and Nurminen; Group difference = -1, 95% CI 2-sided [-3.3 to 1.7]
Statistical Analysis 12: Comparison: MenACWY-CRM + Routine Vaccines vs Routine Vaccines; To demonstrate the non-inferiority of seroresponse to pneumococcal PnC 4 antigen, when PCV is given with MenACWY-CRM, compared with when PCV is given alone; Test type: Non-Inferiority or Equivalence — The immune seroresponse to pneumococcal PnC 4 antigen, when PCV is given concomitantly with MenACWY-CRM, was considered non-inferior to that of PCV given alone, if the lower limit of the two-sided 95% CI for the difference in the percentage of subjects with antibody response was greater than or equal to -10%; Miettinen and Nurminen; Group difference = 1, 95% CI 2-sided [-1.9 to 4.6]
Statistical Analysis 13: Comparison: MenACWY-CRM + Routine Vaccines vs Routine Vaccines; To demonstrate the non-inferiority of seroresponse to pneumococcal PnC 6B antigen, when PCV is given with MenACWY-CRM, compared with when PCV is given alone; Test type: Non-Inferiority or Equivalence — The immune seroresponse to pneumococcal PnC 6B antigen, when PCV is given concomitantly with MenACWY-CRM, was considered non-inferior to that of PCV given alone, if the lower limit of the two-sided 95% CI for the difference in the percentage of subjects with antibody response was greater than or equal to -10%; Miettinen and Nurminen; Group difference = -4, 95% CI 2-sided [-10.3 to 3.2]
Statistical Analysis 14: Comparison: MenACWY-CRM + Routine Vaccines vs Routine Vaccines; To demonstrate the non-inferiority of seroresponse to pneumococcal PnC 9V antigen, when PCV is given with MenACWY-CRM, compared with when PCV is given alone; Test type: Non-Inferiority or Equivalence — The immune seroresponse to pneumococcal PnC 9V antigen, when PCV is given concomitantly with MenACWY-CRM, was considered non-inferior to that of PCV given alone, if the lower limit of the two-sided 95% CI for the difference in the percentage of subjects with antibody response was greater than or equal to -10%; Miettinen and Nurminen; Group difference = -3, 95% CI 2-sided [-8.7 to 2.3]
Statistical Analysis 15: Comparison: MenACWY-CRM + Routine Vaccines vs Routine Vaccines; To demonstrate the non-inferiority of seroresponse to pneumococcal PnC 14 antigen, when PCV is given with MenACWY-CRM, compared with when PCV is given alone; Test type: Non-Inferiority or Equivalence — The immune seroresponse to pneumococcal PnC 14 antigen, when PCV is given concomitantly with MenACWY-CRM, was considered non-inferior to that of PCV given alone, if the lower limit of the two-sided 95% CI for the difference in the percentage of subjects with antibody response was greater than or equal to -10%; Miettinen and Nurminen; Group difference = 0, 95% CI 2-sided [-2.8 to 3.0]
Statistical Analysis 16: Comparison: MenACWY-CRM + Routine Vaccines vs Routine Vaccines; To demonstrate the non-inferiority of seroresponse to pneumococcal PnC 18C antigen, when PCV is given with MenACWY-CRM, compared with when PCV is given alone; Test type: Non-Inferiority or Equivalence — The immune seroresponse to pneumococcal PnC 18C antigen, when PCV is given concomitantly with MenACWY-CRM, was considered non-inferior to that of PCV given alone, if the lower limit of the two-sided 95% CI for the difference in the percentage of subjects with antibody response was greater than or equal to -10%; Miettinen and Nurminen; Group difference = -3, 95% CI 2-sided [-7.3 to 1.6]
Statistical Analysis 17: Comparison: MenACWY-CRM + Routine Vaccines vs Routine Vaccines; To demonstrate the non-inferiority of seroresponse to pneumococcal PnC 19F antigen, when PCV is given with MenACWY-CRM, compared with when PCV is given alone; Test type: Non-Inferiority or Equivalence — The immune seroresponse to pneumococcal PnC 19F antigen, when PCV is given concomitantly with MenACWY-CRM, was considered non-inferior to that of PCV given alone, if the lower limit of the two-sided 95% CI for the difference in the percentage of subjects with antibody response was greater than or equal to -10%; Miettinen and Nurminen; Group difference = 3, 95% CI 2-sided [1.3 to 7.1]
Statistical Analysis 18: Comparison: MenACWY-CRM + Routine Vaccines vs Routine Vaccines; To demonstrate the non-inferiority of seroresponse to pneumococcal PnC 23F antigen, when PCV is given with MenACWY-CRM, compared with when PCV is given alone; Test type: Non-Inferiority or Equivalence — The immune seroresponse to pneumococcal PnC 23F antigen, when PCV is given concomitantly with MenACWY-CRM, was considered non-inferior to that of PCV given alone, if the lower limit of the two-sided 95% CI for the difference in the percentage of subjects with antibody response was greater than or equal to -10%; Miettinen and Nurminen; Group difference = -5, 95% CI 2-sided [-11.4 to 0.5]

6. Secondary Outcome: Geometric Mean Concentrations Of Antibodies Against Routine Concomitant Vaccinations One Month After Infant Series, When Routine Vaccines Are Administered With MenACWY-CRM Compared With When Routine Vaccines Are Given Alone
Description: The immune response was measured as the geometric mean concentrations (GMCs) of antibodies directed against diphtheria, tetanus, pertussis (PT, FHA, Pertactin, FIM), hepatitis B, Hib, polio (type 1, 2 and 3) and pneumococcal (PnC 4, 6B, 9V, 14, 18C, 19F and 23F) antigens when routine vaccines are administered concomitantly with MenACWY-CRM compared with when routine vaccines are given alone, one month after 3 doses of infant series vaccination at 2, 4 and 6 months of age.
Time Frame: One month after third dose of routine infant series vaccination
Population: Analysis was performed on the PP datasets of infants for concomitant, pertussis and hepatitis B vaccinations
Measure: Geometric Mean (95% Confidence Interval); unit: μg/mL
Arm/Group | MenACWY-CRM + Routine Vaccines | Routine Vaccines
Number analyzed (Participants) | 207 | 218
μg/mL
  Diphtheria (N=207,218) | 0.7 [0.63 to 0.78] | 0.85 [0.76 to 0.94]
  Tetanus (N=207,218) | 0.8 [0.7 to 0.91] | 0.67 [0.59 to 0.76]
  PT (N=185,191) | 25 [21 to 30] | 24 [21 to 29]
  FHA (N=185,191) | 48 [43 to 54] | 47 [42 to 52]
  Pertactin (N=185,191) | 56 [47 to 65] | 54 [46 to 62]
  FIM (N=185,191) | 133 [113 to 157] | 122 [105 to 143]
  Polio Type 1 (N=115,113) | 149 [115 to 194] | 117 [89 to 152]
  Polio Type 2 (N=185,179) | 210 [178 to 246] | 185 [156 to 218]
  Polio Type 3 (N=164,162) | 457 [367 to 569] | 402 [321 to 504]
  Hepatitis B (N=138,148) | 394 [284 to 546] | 402 [289 to 558]
  Hib (N=187,194) | 3.75 [2.92 to 4.82] | 2.76 [2.16 to 3.53]
  PnC 4 (N=183,178) | 1.3 [1.16 to 1.46] | 1.45 [1.29 to 1.63]
  PnC 6B (N=183,178) | 1.42 [1.17 to 1.72] | 1.79 [1.47 to 2.18]
  PnC 9V (N=183,178) | 0.95 [0.84 to 1.08] | 1.2 [1.05 to 1.36]
  PnC 14 (N=183,178) | 6.31 [5.45 to 7.31] | 6.61 [5.69 to 7.68]
  PnC 18C (N=183,178) | 1.36 [1.2 to 1.55] | 1.42 [1.24 to 1.62]
  PnC 19F (N=183,178) | 1.84 [1.63 to 2.08] | 2.04 [1.8 to 2.32]
  PnC 23F (N=183,178) | 1.15 [0.99 to 1.35] | 1.33 [1.13 to 1.56]
Statistical Analysis 1: Comparison: MenACWY-CRM + Routine Vaccines vs Routine Vaccines; To demonstrate the non-inferiority of GMC of antibodies to pertussis toxin (PT), when DTaP is given with MenACWY-CRM compared with when DTap is given alone; Test type: Non-Inferiority or Equivalence — The immune response measured as GMC of antibodies to pertussis toxin (PT), when DTaP is given concomitantly with MenACWY-CRM, was considered non-inferior to that of DTaP given alone, if the lower limit of the two-sided 95% CI for the ratio of GMCs (GMC of MenACWY-CRM + Routine Vaccines group divided by GMC of Routine Vaccines group) was greater than 0.67; ANOVA; GMCs ratio = 1.02, 95% CI 2-sided [0.81 to 1.28]
Statistical Analysis 2: Comparison: MenACWY-CRM + Routine Vaccines vs Routine Vaccines; To demonstrate the non-inferiority of GMC of antibodies to pertussis FHA antigen, when DTaP is given with MenACWY-CRM compared with when DTaP is given alone; Test type: Non-Inferiority or Equivalence — The immune response measured as GMC of antibodies to pertussis FHA antigen, when DTaP is given concomitantly with MenACWY-CRM, was considered non-inferior to that of DTaP given alone, if the lower limit of the two-sided 95% CI for the ratio of GMCs (GMC of MenACWY-CRM + Routine Vaccines group divided by GMC of Routine Vaccines group) was greater than 0.67; ANOVA; GMCs ratio = 1.04, 95% CI 2-sided [0.9 to 1.19]
Statistical Analysis 3: Comparison: MenACWY-CRM + Routine Vaccines vs Routine Vaccines; To demonstrate the non-inferiority of GMC of antibodies to pertussis pertactin antigen, when DTaP is given with MenACWY-CRM compared with when DTaP is given alone; Test type: Non-Inferiority or Equivalence — The immune response measured as GMC of antibodies to pertussis pertactin antigen, when DTaP is given concomitantly with MenACWY-CRM, was considered non-inferior to that of DTaP given alone, if the lower limit of the two-sided 95% CI for the ratio of GMCs (GMC of MenACWY-CRM + Routine Vaccines group divided by GMC of Routine Vaccines group) was greater than 0.67; ANOVA; GMCs ratio = 1.04, 95% CI 2-sided [0.84 to 1.28]
Statistical Analysis 4: Comparison: MenACWY-CRM + Routine Vaccines vs Routine Vaccines; To demonstrate the non-inferiority of GMC of antibodies to pertussis FIM antigen, when DTaP is given with MenACWY-CRM compared with when DTaP is given alone; Test type: Non-Inferiority or Equivalence — The immune response measured as GMC of antibodies to pertussis FIM antigen, when DTaP is given concomitantly with MenACWY-CRM, was considered non-inferior to that of DTaP given alone, if the lower limit of the two-sided 95% CI for the ratio of GMCs (GMC of MenACWY-CRM + Routine Vaccines group divided by GMC of Routine Vaccines group) was greater than 0.67; ANOVA; GMCs ratio = 1.09, 95% CI 2-sided [0.88 to 1.35]

7. Secondary Outcome: Geometric Mean Concentrations Of Antibodies Against Pneumococcal Antigens One Month After Toddler Vaccination With PCV Administered With MenACWY-CRM Compared With PCV Given Alone
Description: Immunogenicity was measured as the GMCs of anti-pneumococcal antibodies against pneumococcal antigens PnC 4, 6B, 9V, 14, 18C, 19F and 23F, one month after toddler dose of PCV at 12 months of age administered concomitantly with MenACWY-CRM compared with PCV given alone.
Time Frame: One month after PCV toddler vaccination
Population: Analysis was performed on the PP pneumococcal toddler population.
Measure: Geometric Mean (95% Confidence Interval); unit: μg/mL
Arm/Group | MenACWY-CRM + Routine Vaccines | Routine Vaccines
Number analyzed (Participants) | 161 | 170
μg/mL
  PnC 4 (N=161,170) | 1.57 [1.35 to 1.82] | 1.6 [1.39 to 1.85]
  PnC 6B (N=161,170) | 5.92 [5.05 to 6.95] | 7.8 [6.69 to 9.09]
  PnC 9V (N=161,170) | 1.67 [1.44 to 1.93] | 1.91 [1.66 to 2.19]
  PnC 14 (N=161,170) | 7.9 [6.73 to 9.28] | 7.61 [6.52 to 8.88]
  PnC 18C (N=161,170) | 1.79 [1.55 to 2.08] | 1.8 [1.57 to 2.08]
  PnC 19F (N=161,170) | 5.03 [4.36 to 5.82] | 5.68 [4.95 to 6.53]
  PnC 23F (N=161,170) | 3.3 [2.8 to 3.89] | 3.91 [3.34 to 4.57]
Statistical Analysis 1: Comparison: MenACWY-CRM + Routine Vaccines vs Routine Vaccines; To demonstrate the non-inferiority of GMC of antibodies to pneumococcal PnC 4 antigen when PCV is given with MenACWY-CRM compared with when PCV is given alone; Test type: Non-Inferiority or Equivalence — The immune response as GMC of antibodies to pneumococcal PnC 4 antigen, when PCV is given concomitantly with MenACWY-CRM, was considered non-inferior to that of PCV given alone, if the lower limit of the two-sided 95% CI for the ratio of GMCs (GMC of MenACWY-CRM + Prevnar group divided by GMC of Prevnar group) was greater than 0.50; ANOVA; GMCs ratio = 0.98, 95% CI 2-sided [0.8 to 1.19]
Statistical Analysis 2: Comparison: MenACWY-CRM + Routine Vaccines vs Routine Vaccines; To demonstrate the non-inferiority of GMC of antibodies to pneumococcal PnC 6B antigen when PCV is given with MenACWY-CRM compared with when PCV is given alone; Test type: Non-Inferiority or Equivalence — The immune response as GMC of antibodies to pneumococcal PnC 6B antigen, when PCV is given concomitantly with MenACWY-CRM, was considered non-inferior to that of PCV given alone, if the lower limit of the two-sided 95% CI for the ratio of GMCs (GMC of MenACWY-CRM + Prevnar group divided by GMC of Prevnar group) was greater than 0.50; ANOVA; GMCs ratio = 0.76, 95% CI 2-sided [0.62 to 0.93]
Statistical Analysis 3: Comparison: MenACWY-CRM + Routine Vaccines vs Routine Vaccines; To demonstrate the non-inferiority of GMC of antibodies to pneumococcal PnC 9V antigen when PCV is given with MenACWY-CRM compared with when PCV is given alone; Test type: Non-Inferiority or Equivalence — The immune response as GMC of antibodies to pneumococcal PnC 9V antigen, when PCV is given concomitantly with MenACWY-CRM, was considered non-inferior to that of PCV given alone, if the lower limit of the two-sided 95% CI for the ratio of GMCs (GMC of MenACWY-CRM + Prevnar group divided by GMC of Prevnar group) was greater than 0.50; ANOVA; GMCs ratio = 0.87, 95% CI 2-sided [0.72 to 1.06]
Statistical Analysis 4: Comparison: MenACWY-CRM + Routine Vaccines vs Routine Vaccines; To demonstrate the non-inferiority of GMC of antibodies to pneumococcal PnC 14 antigen when PCV is given with MenACWY-CRM compared with when PCV is given alone; Test type: Non-Inferiority or Equivalence — The immune response as GMC of antibodies to pneumococcal PnC 14 antigen, when PCV is given concomitantly with MenACWY-CRM, was considered non-inferior to that of PCV given alone, if the lower limit of the two-sided 95% CI for the ratio of GMCs (GMC of MenACWY-CRM + Prevnar group divided by GMC of Prevnar group) was greater than 0.50; ANOVA; GMCs ratio = 1.04, 95% CI 2-sided [0.84 to 1.28]
Statistical Analysis 5: Comparison: MenACWY-CRM + Routine Vaccines vs Routine Vaccines; To demonstrate the non-inferiority of GMC of antibodies to pneumococcal PnC 18C antigen when PCV is given with MenACWY-CRM compared with when PCV is given alone; Test type: Non-Inferiority or Equivalence — The immune response as GMC of antibodies to pneumococcal PnC 18C antigen, when PCV is given concomitantly with MenACWY-CRM, was considered non-inferior to that of PCV given alone, if the lower limit of the two-sided 95% CI for the ratio of GMCs (GMC of MenACWY-CRM + Prevnar group divided by GMC of Prevnar group) was greater than 0.50; ANOVA; GMCs ratio = 0.99, 95% CI 2-sided [0.82 to 1.2]
Statistical Analysis 6: Comparison: MenACWY-CRM + Routine Vaccines vs Routine Vaccines; To demonstrate the non-inferiority of GMC of antibodies to pneumococcal PnC 19F antigen when PCV is given with MenACWY-CRM compared with when PCV is given alone; Test type: Non-Inferiority or Equivalence — The immune response as GMC of antibodies to pneumococcal PnC 19F antigen, when PCV is given concomitantly with MenACWY-CRM, was considered non-inferior to that of PCV given alone, if the lower limit of the two-sided 95% CI for the ratio of GMCs (GMC of MenACWY-CRM + Prevnar group divided by GMC of Prevnar group) was greater than 0.50; ANOVA; GMCs ratio = 0.89, 95% CI 2-sided [0.73 to 1.07]
Statistical Analysis 7: Comparison: MenACWY-CRM + Routine Vaccines vs Routine Vaccines; To demonstrate the non-inferiority of GMC of antibodies to pneumococcal PnC 23F antigen when PCV is given with MenACWY-CRM compared with when PCV is given alone; Test type: Non-Inferiority or Equivalence — The immune response as GMC of antibodies to pneumococcal PnC 23F antigen, when PCV is given concomitantly with MenACWY-CRM, was considered non-inferior to that of PCV given alone, if the lower limit of the two-sided 95% CI for the ratio of GMCs (GMC of MenACWY-CRM + Prevnar group divided by GMC of Prevnar group) was greater than 0.50; ANOVA; GMCs ratio = 0.84, 95% CI 2-sided [0.68 to 1.04]

8. Secondary Outcome: Percentage of Subjects With Anti-pneumococcal Antigen Antibodies ≥0.35 μg/mL One Month After Toddler Vaccination With PCV Administered With MenACWY-CRM Compared With PCV Given Alone
Description: The immune seroresponse was measured as the percentage of subjects with anti-pneumococcal antigen antibodies ≥0.35 μg/mL against pneumococcal antigens PnC 4, 6B, 9V, 14, 18C, 19F and 23F, one month after toddler dose of PCV at 12 months of age when administered concomitantly with MenACWY-CRM compared with PCV given alone.
Time Frame: One month after PCV toddler vaccination
Population: Analysis was performed on the PP pneumococcal toddler population.
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | MenACWY-CRM + Routine Vaccines | Routine Vaccines
Number analyzed (Participants) | 161 | 170
Percentage of subjects
  PnC 4 (N=161,170) | 93 [88 to 97] | 96 [92 to 98]
  PnC 6B (N=161,170) | 99 [97 to 100] | 98 [95 to 100]
  PnC 9V (N=161,170) | 97 [93 to 99] | 96 [92 to 98]
  PnC 14 (N=161,170) | 99 [96 to 100] | 99 [97 to 100]
  PnC 18C (N=161,170) | 96 [92 to 99] | 98 [94 to 99]
  PnC 19F (N=161,169) | 99 [96 to 100] | 100 [98 to 100]
  PnC 23F (N=161,170) | 99 [97 to 100] | 98 [94 to 99]

9. Secondary Outcome: Antibody Persistence by Percentage of Subjects With hSBA Titers ≥1:8 Against Serogroup A, C, W and Y, Six Months After Third Infant Vaccination, Prior to MenACWY-CRM Toddler Vaccination
Description: The antibody persistence was measured as the percentage of subjects with hSBA titers ≥1:8 against meningococcal serogroup A, C, W and Y, at baseline and six months after third infant dose of MenACWY-CRM administered at 6 months (12 months of age), before administration of the toddler dose of MenACWY-CRM.
Time Frame: Baseline and Six months after third infant dose of MenACWY-CRM
Population: Analysis was performed on the PP toddler dataset for MenACWY-CRM.
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | MenACWY-CRM + Routine Vaccines | Routine Vaccines
Number analyzed (Participants) | 170 | 178
Percentage of subjects
  Serogroup A - Baseline (N=139, 145) | 1 [0 to 5] | 0 [0 to 3]
  Serogroup A - 6 mo Post-3rd dose (N=168,175) | 7 [4 to 12] | 2 [0 to 5]
  Serogroup C - Baseline (N=126,136) | 7 [3 to 13] | 8 [4 to 14]
  Serogroup C - 6 mo Post-3rd dose (N=156,171) | 37 [30 to 45] | 2 [1 to 6]
  Serogroup W - Baseline (N=152,164) | 15 [9 to 23] | 15 [9 to 23]
  Serogroup W - 6 mo Post-3rd dose (N=153,165) | 70 [62 to 77] | 5 [2 to 9]
  Serogroup Y - Baseline (N=108,113) | 6 [3 to 13] | 5 [2 to 11]
  Serogroup Y - 6 mo Post-3rd dose (N=153,159) | 53 [45 to 61] | 3 [1 to 6]

10. Secondary Outcome: Persistence of hSBA Geometric Mean Titers Against Serogroup A, C, W and Y, Six Months After Third Infant Vaccination, Prior to MenACWY-CRM Toddler Vaccination
Description: The antibody persistence was measured as the hSBA GMTs directed against meningococcal serogroup A, C, W and Y, at baseline and six months after third infant dose of MenACWY-CRM administered at 6 months (12 months of age), before administration of the toddler dose of MenACWY-CRM.
Time Frame: Baseline and Six months after third infant dose of MenACWY-CRM
Population: Analysis was performed on the PP toddler dataset for MenACWY-CRM.
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | MenACWY-CRM + Routine Vaccines | Routine Vaccines
Number analyzed (Participants) | 170 | 178
Titers
  Serogroup A - Baseline (N=139, 145) | 2.07 [1.98 to 2.16] | 2.01 [1.99 to 2.03]
  Serogroup A - 6 mo Post-3rd dose (N=168,175) | 2.52 [2.26 to 2.82] | 2.12 [2.0 to 2.25]
  Serogroup C - Baseline (N=126,136) | 2.49 [2.2 to 2.83] | 2.44 [2.2 to 2.7]
  Serogroup C - 6 mo Post-3rd dose (N=156,171) | 5.98 [4.81 to 7.43] | 2.15 [2.02 to 2.3]
  Serogroup W - Baseline (N=113,126) | 2.99 [2.49 to 3.6] | 2.97 [2.52 to 3.51]
  Serogroup W - 6 mo Post-3rd dose (N=153,165) | 15 [12 to 18] | 2.23 [2.06 to 2.4]
  Serogroup Y - Baseline (N=108,113) | 2.43 [2.19 to 2.71] | 2.32 [2.13 to 2.52]
  Serogroup Y - 6 mo Post-3rd dose (N=153,159) | 8.39 [6.9 to 10] | 2.09 [2.0 to 2.19]

11. Secondary Outcome: Percentage of Subjects With Four-fold Increase in hSBA Titers Against Serogroup A, C, W and Y One Month After Toddler Vaccination of MenACWY-CRM
Description: The immune response was measured as the percentage of subjects who achieved four-fold increase in hSBA titers against meningococcal serogroup A, C, W and Y one month after toddler dose of MenACWY-CRM administered at 12 months of age as compared to hSBA titers before the toddler vaccination.
Time Frame: One month after MenACWY-CRM toddler vaccination
Population: Analysis was performed on the PP toddler dataset for MenACWY-CRM.
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | MenACWY-CRM + Routine Vaccines | Routine Vaccines
Number analyzed (Participants) | 168 | 175
Percentage of subjects
  Serogroup A (N=168,175) | 89 [83 to 93] | 1 [0.014 to 3]
  Serogroup C (N=156,171) | 92 [87 to 96] | 1 [0 to 4]
  Serogroup W (N=153,165) | 95 [91 to 98] | 2 [1 to 6]
  Serogroup Y (N=153,159) | 96 [92 to 99] | 1 [0.016 to 3]

12. Secondary Outcome: Safety of MenACWY-CRM Vaccinations When Administered Concomitantly With Routine Vaccinations
Description: Safety of the study vaccines (MenACWY-CRM and other routine vaccines) was assessed in terms of the number of subjects who reported adverse events (AEs) and/or serious AEs per vaccine group at the following time points: entire study period, after infants vaccination (up to 7 months), between 2- and 4-months, between 4- and 6-months, between 6- and 12-months, between 7- and 12-months, 28 days after 12-month vaccination, and between 29 days after 12-month vaccination and study termination.
  Solicited reactions were not collected during this study. The safety analyses also included any AEs observed by study personnel within 15 minutes following vaccination. All AEs and SAEs were judged by the investigator as whether probably related, possibly related, or not related to vaccine.
Time Frame: From day 1 to 18 months
Population: Analysis was performed on the safety dataset, i.e. all subjects in the exposed population who provided postbaseline safety data
Measure: Number; unit: Number of subjects
Arm/Group | MenACWY-CRM + Routine Vaccines | Routine Vaccines
Number analyzed (Participants) | 255 | 270
Number of subjects
  Entire study - Any AEs | 228 | 239
  Entire study - At least possibly related AEs | 6 | 2
  Entire study - Serious AEs | 21 | 20
  Up to 7 months - Any AEs | 183 | 189
  Up to 7 months - At least possibly related AEs | 6 | 1
  Up to 7 months - Serious AEs | 7 | 8
  Between 2- and 4-months - Any AEs | 99 | 105
  Between 2- & 4-mo - At least possibly related AEs | 1 | 0
  Between 2- and 4-months - Serious AEs | 5 | 5
  Between 4- and 6-months - Any AEs | 118 | 114
  Between 4- & 6-mo - At least possibly related AEs | 3 | 0
  Between 4- and 6-months - Serious AEs | 2 | 2
  Between 6- and 12-months - Any AEs | 187 | 197
  Between 6- & 12-mo - At least possibly related AEs | 2 | 1
  Between 6- and 12-months - Serious AEs | 10 | 2
  Between 7- and 12-months - Any AEs | 175 | 181
  Between 7- & 12-mo - At least possibly related AEs | 0 | 0
  Between 7- and 12-months - Serious AEs | 9 | 2
  28 days post-toddler - Any AEs | 80 | 78
  28 days post-toddler-At least possibly related AEs | 0 | 0
  28 days post-toddler - Serious AEs | 1 | 1
  Between 29 days and study termination - Any AEs | 137 | 137
  B/w 29 days & study terminat-Possibly related AEs | 0 | 0
  Between 29 days and study termination - SeriousAEs | 7 | 11

ADVERSE EVENTS:
Time Frame: Serious adverse events (AEs) were collected throughout the study (from day 1 to 18 months).
Description: Non-serious AEs were also collected throughout the study (from day 1 to 18 months). The number of subjects reported here is from the safety set and not from the enrolled set as reported in the Participant Flow module.
Arm/Group | MenACWY-CRM + Routine Vaccines | Routine Vaccines
Serious Adverse Events (participants affected / at risk) | 21/255 | 20/270
Other Adverse Events (participants affected / at risk) | 216/255 | 227/270
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MenACWY-CRM + Routine Vaccines (N=255) | Routine Vaccines (N=270)
Laryngomalacia (Congenital, familial and genetic disorders) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastrointestinal motility disorder (Gastrointestinal disorders) | 0 (0) | 1 (1)
Impaired gastric emptying (Gastrointestinal disorders) | 1 (1) | 0 (0)
Inguinal Hernia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Abscess (Infections and infestations) | 0 (0) | 2 (2)
Bronchiolitis (Infections and infestations) | 4 (4) | 2 (2)
Cellulitis (Infections and infestations) | 0 (0) | 2 (2)
Clostridial infection (Infections and infestations) | 0 (0) | 1 (1)
Croup infectious (Infections and infestations) | 1 (1) | 3 (3)
Meningitis enteroviral (Infections and infestations) | 1 (1) | 0 (0)
Metapneumovirus infection (Infections and infestations) | 1 (1) | 0 (0)
Otitis media (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 2 (2) | 1 (1)
Pneumonia parainfluenzae viral (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia viral (Infections and infestations) | 1 (1) | 0 (0)
Pyelonephritis (Infections and infestations) | 1 (1) | 1 (1)
Respiratory syncytial virus bronchiolitis (Infections and infestations) | 3 (3) | 2 (2)
Respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1)
Sinusitis (Infections and infestations) | 1 (1) | 0 (0)
Subcutaneous abscess (Infections and infestations) | 1 (1) | 1 (1)
Tonsillitis (Infections and infestations) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 2 (2)
Viral infection (Infections and infestations) | 1 (1) | 0 (0)
Skull fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Moraxella test positive (Investigations) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Failure to thrive (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Cognitive disorder (Nervous system disorders) | 1 (1) | 0 (0)
Convulsion (Nervous system disorders) | 0 (0) | 1 (1)
Febrile convulsion (Nervous system disorders) | 1 (1) | 0 (0)
Hypotonia (Nervous system disorders) | 1 (1) | 0 (0)
Sensory disturbance (Nervous system disorders) | 1 (1) | 0 (0)
Vaginal laceration (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Colectomy (Surgical and medical procedures) | 0 (0) | 1 (1)
Colostomy (Surgical and medical procedures) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MenACWY-CRM + Routine Vaccines (N=255) | Routine Vaccines (N=270)
Conjunctivitis (Eye disorders) | 58 (58) | 52 (52)
Constipation (Gastrointestinal disorders) | 18 (18) | 24 (24)
Diarrhoea (Gastrointestinal disorders) | 25 (25) | 26 (26)
Teething (Gastrointestinal disorders) | 16 (16) | 7 (7)
Vomiting (Gastrointestinal disorders) | 19 (19) | 31 (31)
Pyrexia (General disorders) | 43 (43) | 45 (45)
Bronchiolitis (Infections and infestations) | 37 (37) | 40 (40)
Bronchitis (Infections and infestations) | 15 (15) | 15 (15)
Candida Nappy Rash (Infections and infestations) | 6 (6) | 17 (17)
Candidiasis (Infections and infestations) | 16 (16) | 24 (24)
Croup Infectious (Infections and infestations) | 15 (15) | 21 (21)
Gastroenteritis (Infections and infestations) | 38 (38) | 32 (32)
Otitis media (Infections and infestations) | 100 (100) | 106 (106)
Otitis media acute (Infections and infestations) | 31 (31) | 31 (31)
Pharyngitis (Infections and infestations) | 24 (24) | 32 (32)
Rhinitis (Infections and infestations) | 19 (19) | 20 (20)
Sinusitis (Infections and infestations) | 10 (10) | 15 (15)
Upper respiratory tract infection (Infections and infestations) | 144 (144) | 154 (154)
Viral infection (Infections and infestations) | 36 (36) | 51 (51)
Bronchial Hyperreactivity (Respiratory, thoracic and mediastinal disorders) | 15 (15) | 8 (8)
Cough (Respiratory, thoracic and mediastinal disorders) | 34 (34) | 27 (27)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 17 (17) | 21 (21)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 16 (16) | 8 (8)
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 17 (17) | 17 (17)
Dermatitis diaper (Skin and subcutaneous tissue disorders) | 33 (33) | 40 (40)
Eczema (Skin and subcutaneous tissue disorders) | 29 (29) | 28 (28)
Rash (Skin and subcutaneous tissue disorders) | 13 (13) | 15 (15)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days